CLINICAL TRIAL: NCT00390364
Title: Phase II Study of Single Agent RAD001 in Patients With Colon Cancer and Activating Mutations in the PI3KCA Gene
Brief Title: Everolimus in Treating Patients With Advanced or Metastatic Colorectal Cancer That Did Not Respond to Previous Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawn due to low accrual
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J05107 CDR0000508071; JHOC-J05107; NOVARTIS-JHOC-J05107
Record Dates: First submitted 2006-10-18; First posted 2006-10-19 (Estimated); Results first posted 2014-10-08 (Estimated); Last update posted 2014-10-08 (Estimated); Status verified 2014-10

CONDITIONS: Colorectal Cancer
Keywords: adenocarcinoma of the colon; adenocarcinoma of the rectum; recurrent colon cancer; stage III colon cancer; stage IV colon cancer; recurrent rectal cancer; stage III rectal cancer; stage IV rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Everolimus; Biopsy; Gene Expression Profiling; Immunohistochemistry; Reverse Transcriptase Polymerase Chain Reaction

INTERVENTIONS:
Drug: everolimus
Procedure: antiangiogenesis therapy
Procedure: biopsy
Procedure: diagnostic procedure
Procedure: gene expression analysis
Procedure: immunohistochemistry staining method
Procedure: laboratory biomarker analysis
Procedure: mutation analysis
Procedure: protein tyrosine kinase inhibitor therapy
Procedure: reverse transcriptase-polymerase chain reaction

SUMMARY:
RATIONALE: Everolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

PURPOSE: This phase II trial is studying how well everolimus works in treating patients with advanced or metastatic colorectal cancer that did not respond to previous therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine response rate, time to tumor progression, and survival of patients with advanced or metastatic refractory colorectal cancer and mutations in the PI3K gene treated with everolimus.
* Determine the toxicity profile of this drug in these patients.
* Measure the signaling pathways activated in these patients.
* Determine the pharmacodynamic effects of this drug in these patients.

OUTLINE: This is an open-label study.

Patients receive oral everolimus once daily on days 1-28. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

Patients undergo tumor biopsies and normal skin biopsies at baseline and after the first course of study treatment. Tumor tissue is examined for biological markers (e.g., epidermal growth factor receptor, ERK, Akt, p70s6k, p27, and Rb protein) by immunohistochemistry; apoptosis quantification by TUNEL assay; Ki-67 quantification and Ki-index; gene expression; and c-fos and p27 expression by reverse-transcriptase polymerase chain reaction.

PROJECTED ACCRUAL: A total of 37 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Cytologically or pathologically confirmed colorectal adenocarcinoma

  * Advanced or metastatic disease
* Refractory to ≥ 1 line of prior therapy

  * Not amenable to potentially curative surgical resection
* Mutations in the PI3K gene in tumor tissue
* Tumor tissue available for genetic testing OR willing to undergo baseline tumor biopsy

  * Tumor amenable to sequential biopsies
  * Willing to undergo 2 sequential tumor biopsies, and 2 sequential skin biopsies
* Measurable lesion with ≥ 1 diameter ≥ 2 cm by conventional CT scan (1 cm by spiral CT scan) in a nonirradiated area
* No known brain metastases

PATIENT CHARACTERISTICS:

* ECOG performance status (PS) 0-2 OR Karnofsky PS 60-100%
* Life expectancy > 12 weeks
* WBC ≥ 3,000/mm³
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Bilirubin normal
* AST and ALT ≤ 2.5 times upper limit of normal (ULN)
* Creatinine normal OR creatinine clearance ≥ 60 mL/min
* Cholesterol and triglycerides ≤ 2.5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to everolimus
* No uncontrolled intercurrent illness, including, but not limited to, any of the following:

  * Hypertension
  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness or social situation that would preclude study compliance
* No evidence of bleeding diathesis
* Able to swallow tablets

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy or chemotherapy (6 weeks for nitrosoureas or mitomycin C) and recovered
* No prior targeted therapy against mTOR
* No other concurrent investigational agents
* No concurrent therapeutic anticoagulation

  * Prophylactic anticoagulation (i.e., low-dose warfarin) of venous or arterial access devices allowed provided the requirements for PT, INR or PTT are met.
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent anticancer therapy, including chemotherapy, hormonal therapy, immunotherapy, alternative therapy, or radiotherapy
* No concurrent live vaccination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2006-10; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Hidalgo, MD, PhD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- RAD0001: Eligible patients will be treated with single agent RAD 001 at doses on 10 mg per day orally. Tumor samples will be obtained before and after treatment by means of fine needle aspirate (FNA)-guided tumor biopsies. Treatment effects will be determined by serial MRI scans. Patients will continue treatment until tumor progression or intolerable toxicity.
Period: Overall Study
Arm/Group | RAD0001
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | RAD0001
Number analyzed (Participants) | 1
Age, Continuous [Mean (Full Range); unit: years] | 38 [38 to 38]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Response Rate: The Total Number of Participants With Progression of Disease
Description: To determine response rate and time to tumor progression of patients with colorectal cancer and mutations in the PI3KCA gene who are treated with RAD001. Response and progression will be evaluated in this study using the international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee.
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions assessed by CT (or MRI): Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesion. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesion.
  The outcome measure will be the total number of subjects who show progression of disease.
Time Frame: 1 month
Measure: Number; unit: participants with progression of disease
Arm/Group | RAD0001
Number analyzed (Participants) | 1
participants with progression of disease | 1

ADVERSE EVENTS:
Arm/Group | RAD0001
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RAD0001 (N=1)
headache (General disorders) | 1
sinus infection (Infections and infestations) | 1
rash (Skin and subcutaneous tissue disorders) | 1
hypokalemia (Metabolism and nutrition disorders) | 1
hyperglycemia (Metabolism and nutrition disorders) | 1
leukopenia (Blood and lymphatic system disorders) | 1
thrombocytopenia (Blood and lymphatic system disorders) | 1
lymphopenia (Blood and lymphatic system disorders) | 1
hypercholesterolemia (Metabolism and nutrition disorders) | 1

LIMITATIONS AND CAVEATS:
Out of 28 subjects pre-screened/screened, only one was enrolled and treated, and she progressed after 1 cycle. Study terminated by investigator because of low enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes